CLINICAL TRIAL: NCT01104961
Title: A Masked, Randomized, Prospective, Single Center Crossover Clinical Trial on the Relationship Between Chemically Preserved Contact Lens Packaging Solutions and Bacterial Binding to Corneal Epithelial Cells
Brief Title: Studying the Relationship Between Contact Lens Packaging Solutions and Bacterial Binding to Surface Eye Cells
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Other projects took precedence, no mechanism of funding establed
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Danielle Robertson, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 032010-081
Record Dates: First submitted 2010-04-09; First posted 2010-04-16 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Corneal Ulcer
Keywords: Bacterial infection; Loss of epithelial cells
MeSH Terms: conditions — Corneal Ulcer; Bacterial Infections | interventions — Abortion, Induced

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- Contact Lens Packaging Solution #1 (Experimental): Test solution - contact lens packaging solution
  Interventions: Device: Contact lens packaging solution
- Contact lens packaging solution #2 (Experimental): Test solution - contact lens packaging solution
  Interventions: Device: Contact lens packaging solution
- Balanced salt solution (Placebo Comparator): Control solution
  Interventions: Device: Balanced salt solution (BSS)

INTERVENTIONS:
Device: Contact lens packaging solution — These test solutions are the intervention being tested.
  Other Names: Blister pack solution
  Arms: Contact Lens Packaging Solution #1; Contact lens packaging solution #2
Device: Balanced salt solution (BSS) — BSS is isotonic to the tissues of the eyes.
  Other Names: Saline solution
  Arms: Balanced salt solution

SUMMARY:
The goal of this study is to investigate the overall theory that the use of chemically preserved solutions associated with contact lenses promotes an increase in bacterial infection.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the theory of bacterial binding to surface eye cells through the use of chemically preserved solutions.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 18-38 years
* Any sex, race or national origin accepted as with our past studies. Minority representation will be proactively encouraged.
* No prior history of any contact lens wear within one month of entry into the study.
* No history of allergic eye disease either seasonal or associated with previous contact lens wear.

Exclusion Criteria:

* Any patient that is a current contact lens wearer.
* Patients with active ocular infection or inflammatory disease, history of herpetic keratitis, glaucoma, etc.
* Uncontrolled systemic disease or the presence of any significant illness or condition that could, in the judgment of the investigator, interfere with interpretation of the study results.
* Any patient using ocular tears, anti-histamine based ocular therapies, glaucoma therapy, vasoconstricting drops, etc.

Ages: 18 Years to 38 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-04; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Bacterial binding of Pseudomonas Aeruginosa | 5 weeks
  Counting the number of bacteria that bind to surface epithelial cells.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Robertson, OD, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States